CLINICAL TRIAL: NCT00465270
Title: Randomized Evaluation of Recurrent Stroke Comparing PFO Closure to Established Current Standard of Care Treatment (RESPECT)
Brief Title: Patent Foramen Ovale Closure or Medical Therapy After Stroke - RESPECT Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGA-006; G990318
Expanded Access: NCT00583401 (No longer available)
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Cryptogenic Stroke
Keywords: Cryptogenic; Stroke; PFO; Patent foramen ovale; AMPLATZER; Occluder
MeSH Terms: conditions — Ischemic Stroke; Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Intervention Model Description: AMPLATZER PFO Occluder
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device (Experimental): AMPLATZER PFO Occluder
  Interventions: Device: AMPLATZER PFO Occluder
- Standard or Care - Medical Management (Active Comparator): Medical treatment with Aspirin alone, Coumadin alone, Clopidogrel alone, or Aspirin combined with dipyridamole.
  Interventions: Other: Standard of Care - Medical Management

INTERVENTIONS:
Device: AMPLATZER PFO Occluder — patent foramen ovale closure device
  Arms: Device
Other: Standard of Care - Medical Management — Medical management - aspirin alone, Coumadin alone, Clopidogrel alone, aspirin combined with dipyridamole
  Arms: Standard or Care - Medical Management

SUMMARY:
The purpose of this study is to investigate whether percutaneous Patent Foramen Ovale (PFO) closure, using the AMPLATZER PFO Occluder, is superior to current standard of care medical treatment in the prevention of recurrent embolic stroke.

DETAILED DESCRIPTION:
The AMPLATZER PFO Occluder is a percutaneous, transcatheter occlusion device intended for the non-surgical closure of patent foramen ovale in subjects who have had a cryptogenic stroke due to presumed paradoxical embolism within the last 270 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had a cryptogenic stroke within the last 270 days
* Subjects who have been diagnosed with a Patent Foramen Ovale (PFO)
* Subjects willing to participate in follow-up visits

Exclusion Criteria:

* Subjects with intracardiac thrombus or tumor
* Subjects who have an acute or recent (within 6 months) myocardial infarction or unstable angina
* Subjects with left ventricular aneurysm or akinesis
* Subjects with atrial fibrillation/atrial flutter (chronic or intermittent)
* Subjects with another source of right to left shunt identified at baseline, including an atrial septal defect and/or fenestrated septum
* Subjects with contraindication to aspirin or Clopidogrel therapy
* Pregnant or desire to become pregnant within the next year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 980 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Saver, MD, Principal Investigator — UCLA Stroke Center; John D Carroll, MD, Principal Investigator — University of Colorado, Denver; Richard Smalling, MD, Principal Investigator — University of Texas Houston Health Science Center; David Thaler, MD, Principal Investigator — Tufts Medical Center
Locations (69):
- United States (61):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - LAC + USC Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Summit Medical Center, Oakland, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - University of Colorado, Denver, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Neurologic Associates Inc, Palos Heights, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Southern Illinois University Neurology, Springfield, Illinois
  - Indiana Heart Physicians, Indianapolis, Indiana
  - Ruan Neurology, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Midatlantic Cardiovascular Associates, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Methodist Hospital/Park Nicollet Medical Center, Saint Louis Park, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - University of Medicine and Dentistry of New Jersy, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - DENT Neurologic Institute, Amherst, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Neurology and Neuroscience Associates, Akron, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence St. Vincent's Medical Center, Portland, Oregon
  - Oregon Stroke Center, OHSU, Portland, Oregon
  - LeHigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Milton South Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary's Medical Center, Langhorne, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - St. Thomas Neurology, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical School, Dallas, Texas
  - University of Texas Houston Health Science Center, Houston, Texas
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - UW Medicine Stroke Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - University of Wisconsin Hospital, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Stroke Prevention & Atherosclerosis Research Center (SPARC) - Robarts Research Institute, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Background] Saver JL, Carroll JD, Thaler DE, Smalling RW, MacDonald LA, Marks DS, Tirschwell DL; RESPECT Investigators. Long-Term Outcomes of Patent Foramen Ovale Closure or Medical Therapy after Stroke. N Engl J Med. 2017 Sep 14;377(11):1022-1032. doi: 10.1056/NEJMoa1610057. PMID 28902590
- [Background] Carroll JD, Saver JL, Thaler DE, Smalling RW, Berry S, MacDonald LA, Marks DS, Tirschwell DL; RESPECT Investigators. Closure of patent foramen ovale versus medical therapy after cryptogenic stroke. N Engl J Med. 2013 Mar 21;368(12):1092-100. doi: 10.1056/NEJMoa1301440. PMID 23514286
- See also: Related Info — http://www.respectstudy.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Management: Aspirin alone, Coumadin alone, Clopidogrel alone, or Aspirin combined with dipyridamole.
Period: Overall Study
Arm/Group | Device | Medical Management
Started | 499 | 481
Completed | 395 | 321
Not Completed | 104 | 160
Not completed — Death | 7 | 11
Not completed — Withdrawal by Subject | 34 | 78
Not completed — Lost to Follow-up | 60 | 67
Not completed — Investigator request | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device | Medical Management | Total
Number analyzed (Participants) | 499 | 481 | 980
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (9.7) | 46.2 (10.0) | 45.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 213 | 444
  Male | 268 | 268 | 536

OUTCOME MEASURES:

1. Primary Outcome: Composite of Recurrent Nonfatal Ischemic Stroke, Fatal Ischemic Stroke, or Early Death After Randomization
Description: Nonfatal stroke is defined as: focal neurological deficit presumed to be due to focal ischemia, and either 1) symptoms persisting 24 hours or greater, or 2) symptoms persisting less than 24 hours but associated with MR or CT imaging findings of a new, neuroanatomically relevent, cergral infarct.
  Post-randomization death is defined as: in the MM group as all-cause mortality within 45 days after randomization, and in the device group as all-cause mortality 30 days after implant or 45 days after randomizaiton, whichever occurs last.
Time Frame: Trial enrollment was stopped once 25 unique subjects were mutually adjudicated by the CEC and DSMB as having experienced a primary endpoint event. This occurred on December 20, 2011. The mean follow-up time was 2.6 years.
Population: All primary endpoints that occurred in the trial were recurrent non-fatal ischemic strokes.
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Medical Management
Number analyzed (Participants) | 499 | 481
Participants | 9 | 16
Statistical Analysis 1: Comparison: Device vs Medical Management; Test type: Other; p = 0.08, Log Rank; Cox Proportional Hazard = 0.49, 95% CI 2-sided [0.22 to 1.11]

2. Secondary Outcome: Rate of Complete PFO Closure (Assessed by TEE Bubble Study) at the 6-month Follow-up in the Device Group
Time Frame: 6 months
Population: Only subjects with complete PFO closure data at 6-months were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 349
Participants | 249

3. Post Hoc Outcome: Rate of Recurrent Nonfatal Stroke, Post-randomization Death, and Fatal Ischemic Stroke Through Long Term Follow-up
Time Frame: Long Term Follow-up, median of 5.9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Medical Management
Number analyzed (Participants) | 499 | 481
Participants | 18 | 28
Statistical Analysis 1: Comparison: Device vs Medical Management; Test type: Other; p = 0.046, Log Rank; Cox Proportional Hazard = 0.55, 95% CI 2-sided [0.31 to 0.999]

ADVERSE EVENTS:
Time Frame: The results reported here include adverse events that occurred through the long term follow-up. Patients were followed for a median of 5.9 years.
Arm/Group | Device | Medical Management
All-Cause Mortality (participants affected / at risk) | 7/499 | 11/481
Serious Adverse Events (participants affected / at risk) | 201/499 | 173/481
Other Adverse Events (participants affected / at risk) | 285/499 | 70/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=499) | Medical Management (N=481)
ASD (General disorders) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 2 (2) | 2 (3)
Abnormal Lab Value (General disorders) | 0 (0) | 1 (1)
Acute Bacterial Endocarditis (ABE) (General disorders) | 1 (1) | 0 (0)
Acute Bronchitis (General disorders) | 1 (1) | 0 (0)
Acute Erosive Gastritis (General disorders) | 1 (1) | 0 (0)
Acute Gastroenteritis (General disorders) | 2 (2) | 0 (0)
Acute Pancreatitis (General disorders) | 2 (2) | 0 (0)
Acute Peritonitis (General disorders) | 0 (0) | 1 (1)
Acute Pulmonary Edema (General disorders) | 0 (0) | 1 (1)
Acute Renal Failure (General disorders) | 1 (1) | 1 (1)
Acute Subdural Hematoma (General disorders) | 1 (1) | 0 (0)
Alcohol Intoxication (General disorders) | 1 (1) | 0 (0)
Allergic Device Reaction (General disorders) | 0 (0) | 1 (1)
Allergic Drug Reaction (General disorders) | 2 (2) | 0 (0)
Altered Sensorium (General disorders) | 1 (1) | 0 (0)
Anemias (General disorders) | 4 (4) | 0 (0)
Angina Pectoris (General disorders) | 1 (1) | 1 (1)
Ankle Fracture (General disorders) | 1 (1) | 0 (0)
Anterior Meniscus Tear (General disorders) | 0 (0) | 1 (1)
Anxiety (General disorders) | 0 (0) | 2 (2)
Aortic Aneurysms (General disorders) | 2 (2) | 0 (0)
Appendicitis (General disorders) | 4 (4) | 2 (2)
Arm Fracture (General disorders) | 2 (2) | 1 (1)
Arterial Hypertension/Hypertension (General disorders) | 4 (4) | 1 (1)
Arthritis (General disorders) | 2 (2) | 0 (0)
Asthma (General disorders) | 2 (2) | 1 (1)
Atrial Fibrillation (General disorders) | 6 (8) | 4 (4)
Atrial Flutter (General disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 1 (1) | 2 (2)
Bacterial Infections (General disorders) | 0 (0) | 3 (3)
Bacterial Infections of the Skin (General disorders) | 2 (3) | 1 (1)
Benign Mass (General disorders) | 0 (0) | 1 (1)
Bipolar Disorder (General disorders) | 2 (2) | 0 (0)
Birth Defect (General disorders) | 0 (0) | 1 (1)
Bleeding (General disorders) | 3 (3) | 1 (1)
Blood Loss (General disorders) | 0 (0) | 1 (1)
Bowel Obstruction (General disorders) | 4 (5) | 2 (2)
Brain Abcess (General disorders) | 0 (0) | 1 (1)
Brain Tumor (General disorders) | 0 (0) | 2 (2)
Breast Cancer (General disorders) | 6 (6) | 2 (2)
Bronchiolitis (General disorders) | 0 (0) | 1 (1)
Bronchitis (General disorders) | 0 (0) | 1 (1)
Burns (General disorders) | 1 (1) | 1 (1)
Caesarean Section (General disorders) | 5 (5) | 3 (4)
Cancer (General disorders) | 5 (6) | 7 (7)
Cardiac Arrest (General disorders) | 1 (1) | 3 (3)
Cardiac Perforation (General disorders) | 1 (1) | 0 (0)
Cardiac Thrombus (General disorders) | 2 (2) | 0 (0)
Cardiomyopathy (General disorders) | 1 (1) | 0 (0)
Cellulitis (General disorders) | 2 (3) | 6 (6)
Cerebral Aneurysm (General disorders) | 0 (0) | 2 (2)
Cerebral Infarct - Asymptomatic*** (General disorders) | 0 (0) | 2 (2)
Cerebrospinal Fluid (CSF) Leak (General disorders) | 0 (0) | 1 (1)
Cervical Spondylosis (General disorders) | 1 (1) | 0 (0)
Cervical Stenosis (General disorders) | 2 (2) | 1 (1)
Chest Pain (General disorders) | 18 (19) | 15 (16)
Chest Tightness (General disorders) | 1 (1) | 0 (0)
Chills/Rigors (General disorders) | 1 (1) | 0 (0)
Cholecystitis (General disorders) | 1 (1) | 5 (5)
Choledochal Cysts (General disorders) | 1 (1) | 0 (0)
Choledocholithiaisis (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (General disorders) | 3 (3) | 0 (0)
Chronic Obstructive Airway Disorders (General disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (COPD) (General disorders) | 0 (0) | 1 (1)
Chronic Pancreatitis (General disorders) | 1 (2) | 0 (0)
Closed Head Injury (General disorders) | 1 (1) | 1 (1)
Colitis (General disorders) | 3 (3) | 2 (2)
Colon Cancer (General disorders) | 1 (3) | 1 (1)
Common Cold/Upper Respiratory Tract Infection (General disorders) | 0 (0) | 1 (1)
Compartment Syndrome (General disorders) | 1 (1) | 0 (0)
Complex Partial Seizures (General disorders) | 1 (1) | 0 (0)
Confusion (General disorders) | 0 (0) | 2 (3)
Congestive Heart Failure (General disorders) | 1 (1) | 0 (0)
Conversion Reaction (General disorders) | 2 (3) | 0 (0)
Coronary Artery Disease (General disorders) | 3 (3) | 2 (2)
Cutaneous Abcesses (General disorders) | 2 (2) | 1 (1)
Deep Vein/Venous Thrombosis (General disorders) | 5 (5) | 1 (1)
Dehydration (General disorders) | 0 (0) | 2 (2)
Delirium (General disorders) | 0 (0) | 1 (1)
Depression (General disorders) | 2 (3) | 4 (5)
Disc Protrusion (General disorders) | 1 (1) | 0 (0)
Diverticulitis (General disorders) | 3 (3) | 1 (1)
Dizziness (General disorders) | 2 (3) | 2 (2)
Drug Side Effect (General disorders) | 0 (0) | 1 (1)
Duodenal Cancer (General disorders) | 0 (0) | 1 (1)
Dysarthria/Slurred Speech (General disorders) | 1 (1) | 0 (0)
Dyspnea (General disorders) | 3 (3) | 1 (1)
Elective Surgery (General disorders) | 26 (32) | 17 (20)
Emesis/Vomiting (General disorders) | 0 (0) | 1 (1)
Encephalopathy (General disorders) | 0 (0) | 2 (2)
Eye Lacerations (General disorders) | 0 (0) | 1 (1)
Failure to Thrive (General disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 3 (3) | 2 (2)
Fenestrated Atrial Septum (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Fracture (General disorders) | 3 (4) | 0 (0)
Gastritis (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (General disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (General disorders) | 0 (0) | 2 (2)
Gastrointestinal Bleeding (General disorders) | 6 (6) | 4 (4)
Generalized Seizures (General disorders) | 1 (1) | 1 (1)
Generalized Tonic-Clonic Seizures (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 4 (4) | 1 (1)
Hematoma (General disorders) | 1 (2) | 2 (2)
Hemiparesis/Weakness (General disorders) | 2 (2) | 0 (0)
Hemorrhagic Stroke (General disorders) | 0 (0) | 1 (1)
Hepatic and Biliary Disorders (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Herniated Disc (General disorders) | 2 (2) | 0 (0)
Hip Dislocation (General disorders) | 0 (0) | 1 (2)
Hip Fracture (General disorders) | 1 (1) | 3 (3)
Hip Pain (General disorders) | 0 (0) | 1 (1)
Homicide (General disorders) | 0 (0) | 1 (1)
Hydrocephalus (General disorders) | 1 (1) | 0 (0)
Hypercarbia (General disorders) | 1 (1) | 0 (0)
Hypertensive Encephalopathy (General disorders) | 2 (2) | 1 (1)
Hypoglycemia (General disorders) | 1 (2) | 0 (0)
Hyponatremia (General disorders) | 1 (1) | 0 (0)
Hysterectomy (General disorders) | 5 (5) | 4 (4)
Infective/Bacterial Endocarditis (General disorders) | 1 (1) | 0 (0)
Inferior Myocardial Infarction (General disorders) | 1 (1) | 1 (1)
Inguinal Hernia (General disorders) | 0 (0) | 1 (1)
Intracerebral Haemorrhage (General disorders) | 1 (1) | 0 (0)
Intraparenchymal Haemorrhage (General disorders) | 1 (1) | 1 (1)
Ischemic Eighth Nerve (General disorders) | 1 (1) | 0 (0)
Ischemic Stroke (General disorders) | 18 (19) | 28 (31)
Knee Pain (General disorders) | 1 (1) | 2 (2)
Lacerations (General disorders) | 0 (0) | 1 (1)
Leukemias (General disorders) | 1 (1) | 0 (0)
Long Q-T (General disorders) | 1 (1) | 0 (0)
Low Back Pain (General disorders) | 1 (1) | 0 (0)
Lung Cancer (General disorders) | 1 (1) | 0 (0)
Melanoma (General disorders) | 0 (0) | 1 (1)
Melena (General disorders) | 0 (0) | 1 (1)
Menorrhagia (General disorders) | 1 (1) | 2 (2)
Microcytic Anemia (General disorders) | 1 (1) | 0 (0)
Migraine (General disorders) | 12 (15) | 7 (9)
Missed Abortion (General disorders) | 0 (0) | 2 (2)
Multiple Sclerosis (General disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (General disorders) | 1 (1) | 0 (0)
Myocardial Infarction (General disorders) | 6 (6) | 1 (1)
Nausea (General disorders) | 1 (1) | 0 (0)
Neck Pain (General disorders) | 1 (1) | 0 (0)
Non-Endpoint Transient Ischemic Attack (TIA) (General disorders) | 1 (1) | 0 (0)
Numbness (General disorders) | 3 (3) | 4 (4)
Obesity (General disorders) | 1 (1) | 1 (1)
Orthostatic Hypotension (General disorders) | 1 (1) | 0 (0)
Osler Weber Rendu Syndrome (General disorders) | 0 (0) | 1 (1)
Osteoarthritis/Degenerative Joint Disease (General disorders) | 3 (4) | 6 (7)
Other - Preterm labor (General disorders) | 0 (0) | 1 (1)
Other - SIRS (General disorders) | 1 (1) | 0 (0)
Other - Splenic infarcts (General disorders) | 1 (1) | 0 (0)
Overdose (General disorders) | 4 (7) | 3 (5)
Pain (General disorders) | 1 (1) | 0 (0)
Palpitations (General disorders) | 1 (1) | 1 (1)
Pancreatic Cancer (General disorders) | 0 (0) | 2 (3)
Panic Attack (General disorders) | 1 (1) | 0 (0)
Paresthesia/Paraesthesia (General disorders) | 0 (0) | 1 (1)
Pericardial Effusion (General disorders) | 1 (1) | 1 (1)
Pericardial Tamponade (General disorders) | 2 (2) | 0 (0)
Pericarditis (General disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusion (General disorders) | 1 (1) | 0 (0)
Peripheral Venous Thrombus (General disorders) | 1 (1) | 0 (0)
Pleurisy (General disorders) | 1 (1) | 0 (0)
Pneumonia (General disorders) | 5 (9) | 6 (6)
Pneumonia Caused By Haemophilus Influenzae (General disorders) | 0 (0) | 1 (1)
Pneumothorax (General disorders) | 0 (0) | 1 (1)
Possible Seizure (General disorders) | 2 (2) | 2 (2)
Pre-eclampsia (General disorders) | 0 (0) | 1 (1)
Pregnancy (General disorders) | 2 (2) | 0 (0)
Pregnancy Related Symptoms (General disorders) | 0 (0) | 1 (1)
Premature Ventricular Contraction (General disorders) | 0 (0) | 1 (1)
Presyncope (General disorders) | 0 (0) | 1 (1)
Prostate Discomfort (General disorders) | 1 (1) | 0 (0)
Pulmonary AVM (General disorders) | 2 (2) | 0 (0)
Pulmonary Congestion (General disorders) | 1 (2) | 0 (0)
Pulmonary Embolism (General disorders) | 12 (13) | 3 (3)
Radiculopathy (General disorders) | 0 (0) | 1 (1)
Residual Shunt Requiring Closure (General disorders) | 2 (2) | 0 (0)
Respiratory Illness (General disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (General disorders) | 0 (0) | 1 (1)
Right Hepatic Trocar Injury (General disorders) | 1 (1) | 0 (0)
Rotator Cuff Tear (General disorders) | 0 (0) | 1 (1)
Seizure Disorder (General disorders) | 1 (1) | 1 (1)
Seizure/Convulsions/Epilepsy (General disorders) | 1 (1) | 2 (2)
Sepsis (General disorders) | 4 (8) | 3 (5)
Simple Partial Seizures (General disorders) | 0 (0) | 1 (2)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (General disorders) | 1 (1) | 1 (1)
Spells (General disorders) | 2 (2) | 3 (3)
Spinal Stenosis (General disorders) | 1 (1) | 0 (0)
Spontaneous Abortion (General disorders) | 3 (4) | 1 (1)
Subarachnoid Haemorrhage (General disorders) | 0 (0) | 1 (1)
Subdural Haemorrhage (General disorders) | 0 (0) | 2 (2)
Suicide Attempt (General disorders) | 4 (4) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 3 (3) | 5 (5)
TEE-Related Event (General disorders) | 1 (1) | 0 (0)
Thyroid Cancer (General disorders) | 1 (1) | 1 (1)
Thyroid Disorders (General disorders) | 0 (0) | 1 (1)
Thyrotoxicosis (General disorders) | 0 (0) | 1 (1)
Tingling (General disorders) | 1 (1) | 0 (0)
Transient Global Amnesia (General disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (General disorders) | 8 (8) | 11 (14)
Trauma (General disorders) | 4 (4) | 3 (3)
Tubal Ligation (General disorders) | 1 (1) | 1 (1)
Uncontrolled Blood Sugar (General disorders) | 0 (0) | 1 (1)
Unmasking Old Stroke Symptoms (General disorders) | 3 (3) | 2 (2)
Unstable Angina (General disorders) | 1 (1) | 0 (0)
Unsustained/Nonsustained Ventricular Tachycardia/Cardiac Arrhythmia (General disorders) | 1 (1) | 0 (0)
Urinary Calculi (General disorders) | 2 (2) | 2 (2)
Urinary Incontinence (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infections (General disorders) | 3 (3) | 1 (1)
Uterine Fibroid (General disorders) | 1 (1) | 0 (0)
Uterine Prolapse (General disorders) | 1 (1) | 1 (1)
VASC Bleeding (General disorders) | 2 (2) | 0 (0)
VASC Hematoma (General disorders) | 1 (1) | 0 (0)
Vaginal Child Birth (General disorders) | 10 (10) | 5 (7)
Vaso Vagal Response (General disorders) | 1 (1) | 1 (1)
Vertigo (General disorders) | 5 (5) | 2 (2)
Viral Gastroenteritis (General disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (2) | 0 (0)
Worsening Vision (General disorders) | 0 (0) | 1 (1)
Wound Infection (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=499) | Medical Management (N=481)
Abdominal Pain (General disorders) | 3 (3) | 1 (1)
Abnormal Coagulation Parameter (General disorders) | 0 (0) | 1 (1)
Abnormal Lab Value (General disorders) | 1 (1) | 0 (0)
Acute Erosive Gastritis (General disorders) | 0 (0) | 1 (1)
Acute Pulmonary Edema (General disorders) | 1 (1) | 0 (0)
Allergic Drug Reaction (General disorders) | 7 (7) | 1 (1)
Allergic Dye Reaction (General disorders) | 1 (1) | 0 (0)
Anxiety (General disorders) | 2 (2) | 1 (1)
Asthma (General disorders) | 1 (1) | 0 (0)
Atelectasis (General disorders) | 3 (3) | 0 (0)
Atrial Ectopic Beats/Premature Atrial Beats/Premature Atrial Contractions/Ectopic Atrial Rhythm (General disorders) | 10 (10) | 0 (0)
Atrial Fibrillation (General disorders) | 7 (7) | 0 (0)
Atrial Flutter (General disorders) | 1 (1) | 0 (0)
Atrial Tachycardia (General disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 5 (5) | 0 (0)
Bleeding (General disorders) | 4 (5) | 8 (8)
Borderline Prolongation of QT Interval (General disorders) | 1 (1) | 0 (0)
Bruise/Purpura Simplex (General disorders) | 46 (49) | 26 (28)
Buzzing In Chest (General disorders) | 1 (1) | 0 (0)
Calf Pain (General disorders) | 1 (1) | 0 (0)
Cardiac Thrombus (General disorders) | 1 (1) | 0 (0)
Cellulitis (General disorders) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 47 (48) | 1 (1)
Chest Tightness (General disorders) | 3 (3) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) (General disorders) | 1 (1) | 0 (0)
Contact Dermatitis (General disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 1 (1) | 0 (0)
Couplet (General disorders) | 1 (1) | 0 (0)
Deep Vein/Venous Thrombosis (General disorders) | 1 (1) | 0 (0)
Dental Trauma (General disorders) | 1 (1) | 0 (0)
Device Malposition or Malfunction (General disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 3 (3)
Difficulty Catching Breath (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 4 (4) | 0 (0)
Drug Rash (General disorders) | 2 (2) | 0 (0)
Drug Side Effect (General disorders) | 4 (4) | 5 (5)
Dyspepsia (General disorders) | 1 (1) | 0 (0)
Dyspnea (General disorders) | 7 (7) | 0 (0)
Emesis/Vomiting (General disorders) | 3 (3) | 0 (0)
Epistaxis (General disorders) | 7 (7) | 6 (6)
Esophagitis (General disorders) | 0 (0) | 1 (1)
Fainting/Blackout (General disorders) | 1 (1) | 0 (0)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st degree AV Block (General disorders) | 3 (3) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0)
Gastritis (General disorders) | 3 (3) | 2 (2)
Gastroenteritis (General disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (General disorders) | 1 (1) | 2 (2)
Gastrointestinal Bleeding (General disorders) | 1 (1) | 2 (2)
Gastrointestinal Illness (General disorders) | 1 (1) | 0 (0)
Gingival Bleeding (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 8 (8) | 8 (8)
Heartburn (General disorders) | 2 (2) | 0 (0)
Heaviness of Legs (General disorders) | 1 (1) | 0 (0)
Hematochezia (General disorders) | 0 (0) | 2 (2)
Hematoma (General disorders) | 4 (4) | 2 (2)
Hematuria (General disorders) | 0 (0) | 2 (2)
Hemoptysis (General disorders) | 0 (0) | 1 (1)
Hypotension (General disorders) | 5 (5) | 0 (0)
Hypoxemia (General disorders) | 1 (1) | 0 (0)
Incomplete Right Bundle Branch Block (General disorders) | 3 (3) | 0 (0)
Increased Shunt (General disorders) | 3 (3) | 0 (0)
Instillation Site Foreign Body Sensation (General disorders) | 1 (1) | 0 (0)
Leg Cramps (General disorders) | 1 (1) | 0 (0)
Low Back Pain (General disorders) | 5 (5) | 0 (0)
Low Hematocrit (General disorders) | 1 (1) | 0 (0)
Menorrhagia (General disorders) | 2 (2) | 5 (5)
Meralgia Paraesthetica (General disorders) | 1 (1) | 0 (0)
Mid-Sternal Chest Pressure (General disorders) | 3 (3) | 0 (0)
Migraine (General disorders) | 2 (2) | 0 (0)
Musculoskeletal Pain (General disorders) | 3 (3) | 0 (0)
Nausea (General disorders) | 11 (11) | 0 (0)
Non-Specific EKG Change (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 5 (5) | 0 (0)
Pain Due to a Catheter Drainage Tube (General disorders) | 2 (2) | 0 (0)
Palpitations (General disorders) | 42 (44) | 0 (0)
Paresthesia/Paraesthesia (General disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (General disorders) | 1 (1) | 0 (0)
Paroxysmal Supraventricular Tachycardia (General disorders) | 4 (4) | 0 (0)
Peptic Ulcer Disease (General disorders) | 0 (0) | 1 (1)
Pinching Sensation in Chest (General disorders) | 2 (2) | 0 (0)
Pleural Effusion (General disorders) | 1 (1) | 0 (0)
Post-Menopausal Bleeding (General disorders) | 0 (0) | 1 (1)
Presyncope (General disorders) | 1 (1) | 0 (0)
Pruritus/Itching (General disorders) | 3 (3) | 1 (1)
Pulmonary Congestion (General disorders) | 1 (1) | 0 (0)
Right Axis Deviation (General disorders) | 1 (1) | 0 (0)
Right Bundle Branch Block/Complete Right Bundle Branch Block (General disorders) | 2 (2) | 0 (0)
ST Segment Changes (General disorders) | 1 (1) | 0 (0)
ST-T Wave Abnormality (General disorders) | 3 (3) | 0 (0)
Sick Sinus Syndrome (General disorders) | 1 (1) | 0 (0)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (General disorders) | 19 (20) | 0 (0)
Sinus Tachycardia (General disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 3 (3) | 0 (0)
T-Wave Abnormalities (General disorders) | 1 (1) | 0 (0)
TEE-Related Event (General disorders) | 10 (10) | 1 (1)
Trigeminy (General disorders) | 1 (1) | 0 (0)
Unsustained/Nonsustained Ventricular Tachycardia/Cardiac Arrhythmia (General disorders) | 4 (4) | 0 (0)
VASC Bleeding (General disorders) | 16 (16) | 0 (0)
VASC Bruise (General disorders) | 1 (1) | 0 (0)
VASC Hematoma (General disorders) | 36 (36) | 1 (1)
VASC Pain (General disorders) | 32 (32) | 0 (0)
Vaso Vagal Response (General disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No